CLINICAL TRIAL: NCT01826175
Title: Comparison of Ticagrelor Versus Clopidogrel on Residual Thrombus Burden During Percutaneous Coronary Intervention: an Optical Coherence Tomography Study
Brief Title: Comparison of Ticagrelor Versus Clopidogrel on Residual Thrombus Burden During PCI: an OCT Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated mutually by sponsor & PI due to no enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Ik-Kyung Jang, MD, PhD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2013P000225
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Optical Coherence Tomography; ticagrelor; clopidogrel
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel; Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): Subjects receive 180 mg of ticagrelor immediately prior to coronary artery stenting and have optical coherence tomography imaging after the stenting procedure.
  Interventions: Drug: Ticagrelor; Device: Optical Coherence Tomography
- Clopidogrel (Active Comparator): Subjects receive 600 mg of clopidogrel immediately prior to coronary artery stenting and have optical coherence tomography imaging after the stenting procedure.
  Interventions: Drug: Clopidogrel; Device: Optical Coherence Tomography

INTERVENTIONS:
Drug: Ticagrelor — Subjects are randomized to receive a loading dose of ticagrelor or clopidogrel, and all subjects have Optical Coherence Tomography (OCT) imaging performed at the end of their stenting procedures.
  Other Names: Brilinta; Brilique; Possia
  Arms: Ticagrelor
Drug: Clopidogrel — Subjects are randomized to receive a loading dose of ticagrelor or clopidogrel, and all subjects have Optical Coherence Tomography (OCT) imaging performed at the end of their stenting procedures.
  Other Names: Plavix
  Arms: Clopidogrel
Device: Optical Coherence Tomography — Subjects are randomized to receive a loading dose of ticagrelor or clopidogrel, and all subjects have Optical Coherence Tomography (OCT) imaging performed at the end of their stenting procedures.
  Other Names: OCT

SUMMARY:
Subjects with acute coronary syndromes scheduled for cardiac catheterization will be enrolled in this study. Subjects that are to be treated clinically with coronary artery stenting will be randomized to receive a loading dose of clopidogrel versus ticagrelor after diagnostic angiography but prior to stenting. Optical coherence tomography (OCT) will be performed after stenting and the presence of blood clots inside the new stent will be measured and compared between the groups.

DETAILED DESCRIPTION:
Subjects with acute coronary syndromes scheduled for cardiac catheterization will be enrolled in this study. Subjects that are to be treated clinically with coronary artery stenting will be randomized to receive a loading dose of clopidogrel versus ticagrelor after diagnostic angiography but prior to stenting. Optical coherence tomography (OCT) will be performed after stenting and the presence of blood clots inside the new stent will be measured and compared between the groups

ELIGIBILITY:
Inclusion Criteria:

Patient Characteristics:

1. Males and non-pregnant females > 18 and < 79 years of age presenting with acute coronary syndrome defined as having two of the following criteria:

   1. Signs and symptoms consistent with accelerated angina or prolonged angina (lasting greater than 20 minutes) either at rest or with minimal exertion
   2. ECG changes indicative of new ischemia
   3. Levels of cardiac biomarkers (troponin-T) above the upper limit of the normal range.
2. Patients scheduled to undergo coronary angiography with possible percutaneous coronary intervention (PCI)

Lesion Characteristics on Diagnostic Coronary Angiography

1. De novo lesions in native coronary arteries found by diagnostic coronary angiography
2. Angiographic stenosis <100%
3. Reference vessel diameter 2.5 mm - 4.0 mm by visual estimation

Exclusion Criteria:

General Exclusion Criteria

1. Subjects who are unable or unwilling to sign the informed consent form
2. Subjects being treated with anti-platelet medications other than aspirin prior to diagnostic catheterization including glycoprotein IIb/IIIa inhibitors.
3. Subjects with serious co-morbid conditions that in judgment of the investigator preclude inclusion in this study
4. Subjects with NYHA class III or IV heart failure or known left ventricular ejection fraction < 30%
5. Subjects with an ST elevation myocardial infarction
6. Subjects with hemodynamic or electrical instability (including shock)
7. Subjects diagnosed with severe, non-catheter-related coronary artery spasm
8. Subjects who are or may be pregnant
9. Subjects with known allergies to contrast media
10. Subjects with renal failure as defined by eGFR < 60.
11. History of TIA or stroke < 6 months
12. History of hemorrhagic stroke
13. Hepatic insufficiency defined as liver cirrhosis, AST/ALT/Alkaline Phosphatase greater than 3 times the upper limit of normal or hyperbilirubinemia.

Lesion Specific Exclusion Criteria These exclusion criteria apply to the target lesion to be imaged by OCT.

1. Lesion located in the left main coronary artery
2. Lesions that are heavily calcified
3. Lesions where OCT cannot be performed due to technical difficulties
4. Other lesions that the investigator deems inappropriate for the procedure such as sites with excessive tortuosity or low flow by TIMI grade.
5. Lesion in saphenous vein or arterial conduit

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Total thrombus burden as measured by the volume of in-stent thrombus quantified by planimetry. | Thrombus burden will be measured at the end of the coronary artery stenting procedure.
  The total thrombus burden measured on OCT images will be assessed. The volume of in-stent thrombus will be quantified by planimetry.

SECONDARY OUTCOMES:
PRI (platelet reactivity index) as measured by the PLT-VASP assay. | PRI will be measured at the time of OCT image acquistion (which will occur at the end of the coronary artery stenting procedure).
  The extent of platelet inhibition will be measured by PLT-VASP and VerifyNow P2Y12 assays.
P2Y12 Reaction Units as measured by the VerifyNow P2Y12 assay. | P2Y12 will be measured at the time of OCT image acquistion (which will occur at the end of the coronary artery stenting procedure).
  The extent of platelet inhibition will be measured by PLT-VASP and VerifyNow P2Y12 assays.

OTHER OUTCOMES:
PCI- related myocardial infarction (MI) | PCI-related MI will be assessed within 24 hours after the end of the coronary artery stenting procedure.
  PCI related myocardial infarction is defined by the third Universal defintion of myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Ik-Kyung Jang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No